CLINICAL TRIAL: NCT00111280
Title: HIV-1 Infected Subjects Who Were Randomized in Any Sponsor-selected TMC125 Trial to an Active Control Arm and Either Virologically Failed or Completed the Entire Treatment Period, or to Placebo Arm and Were Treated for at Least 48 Weeks.
Brief Title: TMC125-C211: Trial of TMC125 in HIV-1 Infected Subjects Who Were in a Sponsor Selected TMC125 Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR006742
Record Dates: First submitted 2005-05-18; First posted 2005-05-19 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: HIV Infection
Keywords: HIV infection; TMC125; Nucleoside reverse transcriptase inhibitors (NRTIs); roll-over trial; antiretrovirals (ARVs)
MeSH Terms: conditions — HIV Infections | interventions — etravirine

INTERVENTIONS:
Drug: TMC125

SUMMARY:
This is a Phase II, open-label, roll-over trial to evaluate the long term safety and tolerability of TMC125, administered as part of an individually optimized antiretroviral therapy, in HIV 1 infected subjects. In addition, the antiviral activity and immunological effect of TMC125 as part of an antiretroviral regimen over time, and the evolution of HIV phenotype and genotype will be evaluated.

DETAILED DESCRIPTION:
The purpose of this Phase II, open-label, roll-over trial is to evaluate the long term safety and tolerability of TMC125, administered as part of an individually optimized antiretroviral therapy, in HIV 1 infected subjects. In addition, the antiviral activity and immunological effect of TMC125 as part of an antiretroviral regimen over time, and the evolution of HIV phenotype and genotype will be evaluated. Subjects who were randomized to an active control arm of any sponsor-selected TMC125 trial and virologically failed or completed the entire treatment period, or to placebo arm and were treated for at least 48 and who may derive benefit from TMC125 treatment as judged by the investigator can be enrolled. Based on the currently selected studies, a maximum of 170 subjects will be enrolled in the current trial. A dose of 800mg b.i.d . of TMC125 (formulation TF035) and after the formulation switch, 200mg b.i.d. (formulation F060), will be given in combination with an investigator-selected, optimized underlying therapy starting at baseline and consisting of at least 2 drugs (nucleoside reverse transcriptase inhibitors [NRTIs] and/or allowed protease inhibitors [PIs] and/or enfuvirtide [T 20]) for 48 weeks. Tolerability and safety will be assessed throughout the trial. The efficacy parameters will be determined at defined time points during the trial. The trial will involve a screening visit preferable on the same day as the withdrawal visit of the sponsor-selected trial, a baseline visit, a treatment period of 48 weeks, a final visit and a 4 week follow-up period. TMC125, 800 mg twice a day and after formulation switch, at 200 mg twice a day

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed the Informed Consent Form (ICF) voluntarily
* Male or female subject, aged 18 years and above
* Subject having previously been randomized to an active control arm of a sponsor selected TMC125 trial and has completed the entire treatment period or has met the definition of virological failure, as defined in the original protocol, before TMC125 C211 screening or subjects who were randomized in a fully blinded TMC125 trial, being unblinded after treatment for at least 48 weeks and identified as having received placebo
* Subject agrees to take TMC125 in combination with the investigator-selected combination therapy consisting of at least 2 drugs (NRTIs and/or allowed PI and/or T-20
* low-dose ritonavir [= 400 mg daily dose] is not counted as a separate ARV)
* Subject can comply with the protocol requirements
* Subject's general medical condition, in the investigator's opinion, does not interfere with the assessments and the completion of the trial

Exclusion Criteria:

* History of or currently active alcohol or substance use which in the investigator's opinion would likely compromise the subject's safety or compliance with the study procedures
* Any active clinically significant disease (e.g., tuberculosis, cardiac dysfunction) or findings during physical examination that, in the investigator's opinion, would compromise the subject's safety
* Renal impairment as defined by serum creatinine > 2 x upper limit of normal (ULN)
* Any grade 3 or grade 4 toxicity according to the AIDS Clinical Trial Group (ACTG) grading severity list (except for grade 3 glucose and asymptomatic triglyceride/cholesterol grade 3 or 4 elevations
* or asymptomatic and isolated grade 3 or 4 elevations in gamma-glutamyl transferase [GGT] with all other liver enzymes and bilirubin within normal ranges, or isolated grade 3 elevation in amylase with no increase in lipase and no history of pancreatitis)
* Subjects with clinical or laboratory evidence of significantly decreased hepatic function or decompensation, irrespective of liver enzyme levels (International Normalized Ratio > 1.3 or albumin < 30 g/l or direct bilirubin > 2.5 x ULN).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-09; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of the trial is to evaluate the long-term safety and tolerability of TMC125.

SECONDARY OUTCOMES:
The secondary objectives are to evaluate the antiviral activity and immunological effect of TMC125 as part of an antiretroviral (ARV) regimen over time, and to evaluate genotypic and phenotypic changes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- See also: Clinical Study Report Synopsis of TMC125-C211: Trial of TMC125 in HIV-1 Infected Subjects Who Were in a Sponsor Selected TMC125 Trial. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=995&filename=CR006742_CSR.pdf